CLINICAL TRIAL: NCT04641689
Title: Stand Up Kansas: An Intervention to Reduce Sedentary Behavior in the Workplace
Brief Title: Stand Up Kansas: An Intervention to Reduce Sedentary Behavior in the Home Work Environment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kansas State University (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Emily Mailey, Associate Professor, Kansas State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB8886
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Sedentary Behavior; Behavior, Health; Cholesterolemia; Obesity; Stress; Hypertension; Fatigue; Glucose, High Blood; Mood
Keywords: physical activity
MeSH Terms: conditions — Sedentary Behavior; Health Behavior; Obesity; Hypertension; Fatigue; Motor Activity

STUDY DESIGN:
Intervention Model Description: 2 x 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Desk Only (Active Comparator): Participants will receive a height-adjustable desk to use in their home work environment.
  Interventions: Device: Desk Only
- Program Only (Active Comparator): Participants will receive 12 weeks of online content to support reductions in sedentary behavior while working from home. Content will be based on social cognitive theory.
  Interventions: Behavioral: Program Only
- Desk + Program (Experimental): Participants will receive a height-adjustable desk to use in their home work environment AND 12 weeks of online content to support reductions in sedentary behavior while working from home.
  Interventions: Device: Desk Only; Behavioral: Program Only
- Waitlist Control (No Intervention): Participants will receive the intervention (desk + program) after all follow-up data have been collected.

INTERVENTIONS:
Device: Desk Only — Provision of height-adjustable desk
  Other Names: VariDesk Pro Plus 36 height-adjustable desk
  Arms: Desk + Program; Desk Only
Behavioral: Program Only — Online modules will promote goal setting, self-monitoring, habit formation, social support, barrier identification, and environmental modifications
  Arms: Desk + Program; Program Only

SUMMARY:
This project will examine the effectiveness of an intervention to reduce sedentary behavior in Kansas State University employees who are primarily working from home. We will recruit 100 employees to participate. Participants will be randomly assigned to one of four conditions: desk only, program only, desk + program, or waitlist control. The program will consist of strategies to reduce sitting and increase physical activity in the home environment. We will assess whether the intervention successfully elicits reductions in sitting among employees, as well as changes in cardiometabolic and work-related outcomes.

DETAILED DESCRIPTION:
For this project we will conduct a 12-week intervention that incorporates multiple strategies to reduce sedentary behavior among university employees who are primarily working from home. Participants will be recruited via campus networks.

Participants will attend an initial testing visit, during which anthropometric and health outcome data (blood pressure, blood glucose and cholesterol) will be collected. Following the testing visit, all participants will complete an activity log for the next 5 work days, and a subsample will wear an activPAL 4 device for 7 days. All participants will complete a series of questionnaires (measuring physical activity, fatigue, stress, productivity, mood, and diet) online.

After all baseline data have been collected, participants will be randomized to one of four conditions: desk only, program only, desk + program, or waitlist control. Those in the desk only and desk+program conditions will receive a height-adjustable desk. They will be asked to set up the desk at their home workstation and send a photo of the setup to our research team within one week. Those in the program only and control conditions will receive their height-adjustable desks after completing the post-intervention assessments. Participants assigned to the program only and desk+program conditions will have access to a website that includes a variety of resources for reducing sedentary behavior and increasing physical activity in the home environment. The intervention program will be based on social cognitive theory and will be designed to promote self-efficacy, self-regulation, positive outcome expectations, and social and environmental support. Participants will complete weekly modules that include activities such as goal setting and self-monitoring, action and coping planning, group discussions, etc. The program will also provide suggestions for changes to the home work environment, access to virtual stretching and strengthening videos, examples of technology to prompt breaks, etc. Participants will also receive 2 small group coaching calls via Zoom (at 3 and 8 weeks) to assist them in setting goals for reducing sedentary behavior and overcoming barriers. Participants in the desk only and waitlist control groups will receive access to the program after completing the post-intervention assessments.

All measures will be repeated following the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employee (works >30 hours per week)
* Sedentary job (>75% of workday seated)
* Working primarily at home (>80% of typical week)
* Able to safely engage in light intensity physical activity
* No ambulatory limitations

Exclusion Criteria:

* Working <30 hours per week
* Standing or physically active >25% of typical workday
* Working on campus >20% of a typical week OR planning to resume work on campus in the next 3 months
* Uncontrolled stage 2 (severe) hypertension without a medical release signed by a physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change in sedentary behavior during the workday | Baseline and 12 weeks
  Measured via 5-day activity log

SECONDARY OUTCOMES:
Change in physical activity | Baseline and 12 weeks
  International Physical Activity Questionnaire (long form)
Changes in sitting, standing and stepping | Baseline and 12 weeks
  activPAL (subsample)
Change in productivity | Baseline and 12 weeks
  Health and Work Questionnaire
Change in stress | Baseline and 12 weeks
  Perceived Stress Scale (4-item)
Change in fatigue | Baseline and 12 weeks
  Fatigue Symptom Inventory
Change in mood | Baseline and 12 weeks
  Positive and Negative Affect Schedule
Change in diet | Baseline and 12 weeks
  Rapid Eating Assessment for Participants - Shortened Version
Change in blood pressure | Baseline and 12 weeks
  Measured using automatic blood pressure cuff
Change in fasting blood glucose | Baseline and 12 weeks
  Blood sample obtained via finger stick
Change in cholesterol | Baseline and 12 weeks
  Total, HDL, and LDL; Blood sample obtained via finger stick
Change in triglycerides | Baseline and 12 weeks
  Blood sample obtained via finger stick
Change in waist circumference | Baseline and 12 weeks
  Measured to the nearest 0.5 cm
Change in weight | Baseline and 12 weeks
  Measured in kg

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Mailey, PhD, Principal Investigator — Kansas State University
Locations (1):
- Kansas State University, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT04641689/ICF_000.pdf